CLINICAL TRIAL: NCT01141595
Title: Biomarkers of Central Nervous System Tetrahydrobiopterin Concentration and Response to Tetrahydrobiopterin Supplementation in Children With Idiopathic Cognitive Developmental Disorders
Brief Title: Tetrahydrobiopterin Treatment in Children With Idiopathic Cognitive Developmental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Richard Frye, Associate Professor of Pediatrics, Directory of Autism Research, Arkansas Children's Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-09-0578
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kuvan® (Experimental): Patients will be instructed to take 20 mg/kg/day of Kuvan® orally dissolved in 4 - 8oz. of water or apple juice with breakfast.
  Interventions: Drug: sapropterin dihydrochloride

INTERVENTIONS:
Drug: sapropterin dihydrochloride — Patients will be instructed to take 20 mg/kg/day of Kuvan® orally dissolved in 4 - 8oz. of water or apple juice with breakfast.
  Other Names: Kuvan®

SUMMARY:
The purpose of this study is to develop biomarkers for central nervous system BH4 concentration in children with autism so they can be easily screened to determine if they may benefit from BH4 supplementation. Kuvan is a synthetic form of BH4. BH4 is an enzyme cofactor that is essential for several critical metabolic functions.

DETAILED DESCRIPTION:
SUMMARY

PURPOSE: The purpose of this study is to develop biomarkers for central nervous system BH4 concentration in children with autism so they can be easily screened to determine if they may benefit from BH4 supplementation. Kuvan is a synthetic form of BH4. BH4 is an enzyme cofactor that is essential for several critical metabolic functions.

Procedures: Consented subjects' behavior, particularly irritability, cognitive and language function will be assessed at baseline to make sure that the subject meets the inclusion and exclusion criteria. Parents of subjects will be instructed to give the subjects 20 mg/kg/day of Kuvan® orally dissolved in 4 - 8oz. of water or apple juice with breakfast. Subjects will not be permitted to start any new supplement treatments during the study period but will be allowed to continue previous supplements. Subjects will be permitted to take over the counter medications or other prescription medications for acute illnesses. Evaluation of subjects will include three clinic visits for neuropsychological and clinical testing, completion of study-related questionnaires and telephone follow-up visits.

Course of Study: Subjects will be in the study for up to 16 weeks.

Enrollment: The study will enroll 20 (male and female) subjects, 2-6 years old, with delays in language and/or social development. Vulnerable populations include children. A pediatric risk assessment was completed by Ian Butler, MD with an outcome of minimum risks to subjects.

Recruitment: Subjects will be recruited when their parents present them for care at the University of Texas medically-based autism clinic.

Known Risks: For the study drug Kuvan, there have been rare associations with gastroesophageal reflux and a previous form of this compound was associated with seizures in individuals taking Levodopa concurrently. There is a risk of loss of confidentiality.

Data Safety Monitoring: A DSMB will not be formed for this study. The PI will be responsible for the data and safety of the study.

Informed Consent: A written parental informed consent form has been submitted for review and approval. There is no cost for participation, and no remuneration. Confidentiality will be maintained through the use of unique study codes.

IND#: A request for a pre-IND meeting with the FDA to discuss the possible IND exemption has been submitted.

Funding Source: This study is being funded by BioMarin Pharmaceuticals.

SCIENTIFIC PRE-REVIEW: The Clinical Research Unit Review Board Committee Scientific Advisory Committee (SAC) completed the submission with the outcome of CRU - Approved on12/10/2009.

ELIGIBILITY:
Inclusion Criteria:

1. Children 2 years 0 months to 6 years 11 months of age will be recruited.
2. Delay in language and/or social development with or without delays in gross and/or fine motor development.
3. CSF BH4 level less than or equal to 30 nM/L as determined by lumbar puncture.
4. Adaptive Behavior greater than 50 as determined by the Vineland Adaptive Behavior Scale.

Exclusion Criteria:

1. Epilepsy / Seizure disorder as determined by medical history.
2. Epileptiform discharges without clinical seizures.
3. Metabolic disorder that would be a contraindication to tetrahydrobiopterin treatment.
4. Genetic disorder
5. Therapies that cannot be maintained at a constant level or have not been ongoing for more than 3 months as determined by medical history
6. Prematurity
7. Developmental delay isolated to motor delay.
8. Current gastroesophageal reflux
9. Current or history of liver or kidney disease
10. Severe irritability (as determined by the aberrant behavior checklist)
11. Drugs known to affect folate metabolism (e.g., methotrexate) and their derivatives
12. Patients who are receiving drugs that affect nitric oxide-mediated vasorelaxation (e.g., PDE-5 inhibitors such as sildenafil, vardenafil, or tadalafil)
13. Patients who are receiving levodopa.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Frye RE, Huffman LC, Elliott GR. Tetrahydrobiopterin as a novel therapeutic intervention for autism. Neurotherapeutics. 2010 Jul;7(3):241-9. doi: 10.1016/j.nurt.2010.05.004. PMID 20643376
- [Background] Frye RE. Central tetrahydrobiopterin concentration in neurodevelopmental disorders. Front Neurosci. 2010 Jul 8;4:52. doi: 10.3389/fnins.2010.00052. eCollection 2010. PMID 20661295
- [Result] Frye RE, DeLatorre R, Taylor HB, Slattery J, Melnyk S, Chowdhury N, James SJ. Metabolic effects of sapropterin treatment in autism spectrum disorder: a preliminary study. Transl Psychiatry. 2013 Mar 5;3(3):e237. doi: 10.1038/tp.2013.14. PMID 23462988
- See also: Manuscript of Study Results — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3625913/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited from a medical clinic specalizing in neurodevelopmental disorders
Pre-assignment Details: No significant events
Period: Overall Study
Arm/Group | Kuvan®
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Kuvan®
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.0 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Preschool Language Scales
Description: Change in the raw score from baseline of the Preschool Language Scales over the 16 week period. The raw score was measured at baseline, 8 weeks and 16 weeks after starting treatment and the change over the 16 week period from baseline to the end of the study was calculated. There was no imputed data and the analysis was as treated. The raw score ranged from 0 to 130. Higher scores indicate better performance.
Time Frame: 16 weeks
Population: The number of participants with data available that completed at least the 16 week assessment.
Measure: Mean (Standard Deviation); unit: Raw score units / 16 weeks
Arm/Group | Kuvan®
Number analyzed (Participants) | 8
Raw score units / 16 weeks | 7.6 (8.4)

ADVERSE EVENTS:
Arm/Group | Kuvan®
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kuvan® (N=10)
Irritability (Psychiatric disorders) | 1 (1)
Excitement (Psychiatric disorders) | 1 (1)
Upset stomach (Gastrointestinal disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No